CLINICAL TRIAL: NCT03365336
Title: Indian Herbal Medicine for Influenza - Randomized Controlled Study
Brief Title: Influenza Management With Polyherbal Formulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Composite Interceptive Med Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OI-008-2017
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Intervention Model Description: Parallel follow up of two groups randomly allocated through a central randomization process.
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Each Flu Care capsule consists of combination of seven polyherbal formulation (350 mg). Participant will be instructed to take one capsule thrice daily at a fixed time in the day for the study duration of 7 days along with 75 mg of Oseltamivir.
  Interventions: Drug: polyherbal formulation; Drug: Oseltamivir 75mg
- Standard Care Group (Active Comparator): Standard of care consist of 75 mg of Oseltamivir for five days and any other required provision of care. These will be determined on case by case basis by research clinician.
  Interventions: Drug: Oseltamivir 75mg

INTERVENTIONS:
Drug: polyherbal formulation — Each Flu Care consist of 350 mg of polyherbal component
  Other Names: Flu Care
  Arms: Intervention Group
Drug: Oseltamivir 75mg — All the participant has to take 75 mg of oseltamivir for five days.

SUMMARY:
The aim of this study is to determine the efficacy of Flu care polyherbal formulation in the management of acute uncomplicated case of Influenza within 48 hours of symptoms onset.

DETAILED DESCRIPTION:
Influenza is one of the most common epidemics occurring in India during winter months. Most of the commonly used antiviral have limited efficacy and safety in influenza treatment. Flu Care polyherbal consist of antiviral, antitussive and anti-inflammatory herbal medicine. If this Flu care intervention is shown to be effective, there will be major potential benefits to general population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects above the age of 18 years, providing written informed consent.
* Patients with a duration of influenza symptoms confirmed by all of the following:

  1. Fever ≥ 38º C (axillary) during the predose examinations or within the 4 hours prior if antipyretics were taken
  2. At least 1 each of the following general and respiratory symptoms associated with influenza is present with a severity of moderate or greater: i. General symptoms (headache, feverishness or chills, muscle or joint pain, or fatigue) ii. Respiratory symptoms (cough, sore throat, or nasal congestion) Rapid diagnostic test, PCR, or viral culture positive for influenza in the 96 hours prior to first dose
* The time interval between the onset of symptoms and the predose examinations is 48 hours or less. The onset of symptoms is defined as either:

  1. Time of the first increase in body temperature (an increase of at least 1º C from normal body temperature)
  2. Time when the patient experiences at least 1 new general or respiratory symptom

Exclusion Criteria:

Patients will be considered at high risk of influenza complications due to the presence of at least 1 of the following inclusion criteria:

1. Asthma or chronic lung disease (such as chronic obstructive pulmonary disease or cystic fibrosis)
2. Endocrine disorders (including diabetes mellitus)
3. Residents of long-term care facilities (e.g., nursing homes)
4. Compromised immune system (including patients receiving corticosteroids not exceeding 20 mg of prednisolone or equivalent, and patients being treated for human immunodeficiency virus (HIV) infection with a cluster of differentiation 4 count > 350 cells/mm³ within the last 6 months)
5. Neurological and neurodevelopmental disorders (including disorders of the brain, spinal cord, peripheral nerve, and muscle, e.g., cerebral palsy, epilepsy [seizure disorders], stroke, muscular dystrophy, or spinal cord injury)
6. Heart disease (such as congenital heart disease, congestive heart failure, or coronary artery disease), excluding hypertension without any other heart-related symptoms
7. Adults aged ≥ 65 years
8. Blood disorders (such as sickle cell disease)
9. Metabolic disorders (such as inherited metabolic disorders and mitochondrial disorders)
10. Morbid obesity (body mass index ≥ 40)

Other Exclusion criteria Any one of the following

* Influenza vaccination with live attenuated vaccine in the 3 months prior to randomization
* Antiviral treatment for influenza in 2 weeks prior to randomization
* Severe Hepatic and renal impairment
* Pregnant, attempting to conceive, or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-15 (Estimated); Study Completion 2018-05-15 (Estimated)

PRIMARY OUTCOMES:
Time to improvement of symptoms | Day 1 pretreatment upto Day 7
  Time to improvement of symptoms is defined as the time from initiation of study treatment to improvement of influenza symptoms for a duration of at least 21.5 hours (24 hours - 10%).

SECONDARY OUTCOMES:
Percentage change in participants positive for influenza virus titer and viral RNA at end of treatment | 7 days
  Defined as the percentage of patients whose virus titer and ribonucleic acid (RNA) load are become less than the lower limit of quantification among those assessed for virus titer and RNA load. RNA load is measured by reverse transcription polymerase chain reaction (RT-PCR).
Time to alleviation of symptoms | Day 1 pretreatment up to Day 7
  Time to alleviation of symptoms is defined as the time between the initiation of the study treatment and the alleviation of influenza symptoms. The alleviation of influenza symptoms is defined as the time when all of 7 influenza symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) have been assessed by the patient.
Time to improvement in the 4 systemic symptoms | Day 1 pretreatment up to Day 7
  Defined as the time between the initiation of the study treatment and the improvement in the 4 systemic symptoms symptoms (headache, feverishness or chills, muscle or joint pain, and fatigue).
Time to improvement in the 3 respiratory symptoms | Day 1 pretreatment up to Day 7
  Defined as the time between the initiation of the study treatment and the improvement in the 3 respiratory symptoms (cough, sore throat, and nasal congestion).
Time to resolution of fever | Day 1 pretreatment up to Day 7
  Defined as the time between the initiation of the study treatment and the resolution of fever.
  The resolution of fever is defined as the time when the patient's self-measured temperature becomes less than 37º C.
Percentage of participants with adverse events | Baseline up to Day 7
Percentage of participants who had been hospitalized | Baseline up to Day 7
Percentage of participants with influenza-related complications | Baseline up to Day 7
  Defined as the percentage of patients who experience each influenza-related complication (hospitalization, death, sinusitis, otitis media, bronchitis, and radiologically-confirmed pneumonia) as an adverse event after the initiation of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dayanand B Yaligar, MBBS, Principal Investigator — Narayana Hrudayalaya Hospital
Locations (1):
- Mazumdar Shaw Medical Centre, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided